CLINICAL TRIAL: NCT05676593
Title: Interest of Freestyle Libre 2 as a Tool for Therapeutic Education in Recently Diagnosed Type 2 Diabetics Patients
Brief Title: Interest of FSL 2 in Recently Diagnosed Type 2 Diabetic Patients
Acronym: FREEDIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL22_0232
Record Dates: First submitted 2022-12-06; First posted 2023-01-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Endocrinology; Type 2 Diabetes
Keywords: Sensor; Therapeutic education; Diabete; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: We therefore propose a prospective randomised study in 2 arms :
  * a group of people living with diabetes receiving standard TPE vs
  * a group of people living with diabetes receiving standard TPE + FSL 28 days Ourmain objective is to determine the benefit of CGM on HbA1c at 3 months between 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People living with diabete standard TPE (Active Comparator): HBA1c at 3 and 6 months Therapeutic education Auto questionnary on Aviitam plateform at 3 and 6 months
  Interventions: Other: Therapeutic education
- People living with diabete standard TPE + FSL 28 days (Experimental): Continuous mesure of glucose (FSL2) during 28 days at enrollment Therapeutic education HBA1c at 3 and 6 months Auto questionnary on Aviitam plateform at 3 and 6 months
  Auto questionnary on Aviitam plateform at 3 and 6 months
  Interventions: Device: Freestyle Libre 2; Other: Therapeutic education

INTERVENTIONS:
Device: Freestyle Libre 2 — The FSL will be placed on patient for 28 days to measure interstitial glucose
  Arms: People living with diabete standard TPE + FSL 28 days
Other: Therapeutic education — Therapeutic education

SUMMARY:
Therapeutic patient education (TPE) is a key element in the management of people living with type 2 diabetes.

The benefit of therapeutic education (TPE) has been clearly established on glycaemic control.

Continuous interstitial glucose monitoring (CGM) can be considered as a TPE tool for people living with diabetes. A direct reading of the effects of diet and physical activity on glycaemic levels could have an impact on the initiation and maintenance of therapeutic lifestyle modifications.

The investigators therefore propose a prospective randomised study in 2 arms :

* a group of people living with diabetes receiving standard TPE vs
* a group of people living with diabetes receiving standard TPE + FSL 28 days Ourmain objective is to determine the benefit of CGM on HbA1c at 3 months between 2 arms

DETAILED DESCRIPTION:
Main objective to the investigators is to determine the benefit of continuous interstitial glucose monitoring (by fresstyle 2) for 28 days coupled with standard TPE (Patient Therapeutic Education) vs standard TPE alone in newly diagnosed type 2 diabetics on HbA1c at 3 months.

The secondary objectives are to evaluate the effect of the TPE coupled with FSL vs TPE alone on :

* HbA1c at 6 months (assessment of persistence or not of a remote effect)
* weight change at 3 and 6 months
* other cardiovascular risk factors : variation in blood pressure, lipid profil at 3 and 6 months
* eating behaviour/ eating habits at 3 and 6 months
* treatment satisfaction, anxiety and quality of life scores

ELIGIBILITY:
Inclusion Criteria:

* recently diagnosed diabete mellitus (<1 an) treated by non medical therapeutics and/or metformine
* > 18 years old
* initial glycated hemoglobin between 7 and 8.5%

Exclusion Criteria:

* Person whose physical and/or psychological health is severely impaired
* Person deprived of his rights, person under guardianship or curatorship
* Person deprived of liberty (by judicial or administrative decision)
* Person who does not speak the French language
* Absence of affiliation to/Not beneficiary of a Social Security scheme
* Absence of written informed consent to participate in the study
* Unable to understand the nature, purpose and methodology of the study
* Bariatric surgery planned within 6 months of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-11-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Rate of change in glycated hemoglobine at 3 months | 3 months
  biological control of glycated hemoglobin in a laboratory

SECONDARY OUTCOMES:
Rate of change of the time in range, time above range and time below range | 6 months
  data of the freestyle libre
Rate of change in glycated hemoglobin at 6 months | 6 months
  biological control
Rate of change in weight in kg | In kg each 3,6 months
Quality of Life questionnary | Set a score out of 100 (100 good good quality of life - 0 bad quality of life) performed at 3,6 months
  EQVOD - Scale of Quality of Life, Obesity and Dietetics
Rate of change arteriel pressure | In mmHg each 3,6 months
Concentration of of LDL cholesterol | In g/L each 3,6 months
Concentration of Triglyceride | In g/L each 3,6 months
Anxiety and depression scale questionnary | 14 questions (high score depression, anxiety - low score good health) performed at 3,6 months
  HAD - Hospital Anxiety and Depression scale
Quality of Life questionnary | From 0 to 100 (100 good quality of life - 0 bad quality of life) performed at 3,6 months
  EQ-5D - EuroQoL-5D
Eating behavior questionnaire | 33 questions (no scale, doctor's assessment of the answers) performed at 3,6 months
  DEBQ-Dutch Eating Behaviour Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UHM Montpellier, Montpellier, France